CLINICAL TRIAL: NCT01418820
Title: Paraorbital-Occipital Alternating Current Stimulation Therapy of Patients With Post-Chiasmatic Lesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Magdeburg (Other)
Collaborators: EBS Technologies GmbH (Industry)
Responsible Party: Principal Investigator, Bernhard A. Sabel, Prof. Dr., University of Magdeburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EBS-PP-2011-02-16-001
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Complete Hemianopia; Incomplete Hemianopia; Scotoma; Quadrantanopia; Stroke; Hemorrhage; Brain Trauma
Keywords: hemianopia; visual field defect; stroke; non-invasive brain stimulation; alternating current stimulation
MeSH Terms: conditions — Scotoma; Hemianopsia; Stroke; Hemorrhage; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum stimulation (Experimental): repetitive transorbital alternating current stimulation (rtACS)
  Interventions: Device: Verum stimulation
- Placebo stimulation (Sham Comparator): compared to verum stimulation the same electrode montage set-up is used during placebo stimulation, except that placebo patients receive a minimal stimulation
  Interventions: Device: Placebo stimulation

INTERVENTIONS:
Device: Verum stimulation — 10 days (2x 5 working days), daily transorbital alternating current stimulation (rtACS) is applied with a device generating weak current pulses in predetermined firing bursts of 2 to 9 pulses. The amplitude of each current pulse is below 1000 µA. Current intensity is individually adjusted according to how well patients perceived phosphenes, e.g. any sensation of flickering light in response to the rtACS stimulation. Stimulation frequencies were between the individual alpha frequency peak and below flicker fusion.
  Arms: Verum stimulation
Device: Placebo stimulation — 10 days (2x 5 working days), daily sham-stimulation with the same electrode montage set-up that is used for verum transorbital alternating current stimulation (rtACS). Minimal sham-stimulation was performed with single bursts (approx. one per min) of electrical currents at a given frequency of 5Hz and individually adjusted current amplitude.
  Arms: Placebo stimulation

SUMMARY:
Visual field areas, which are not absolutely blind, are hypothesized to have some residual capacities that constitute their potential for vision restoration. Vision restoration can be achieved by varies methods including behavioral training and electrical brain stimulation such as transcranial direct current stimulation (tDCS) and repetitive transorbital alternating current stimulation (rtACS) which are able to influence the excitability and activity of cortical areas.

It is hypothesized that transorbital alternating current stimulation (tACS) can improve the residual field of vision in patients with post-chiasmatic lesions.

ELIGIBILITY:
Inclusion Criteria:

* lesion of the tractus opticus or of the visual cortex
* lesion age > 6 months
* stable visual field defect with residual vision

Exclusion Criteria:

* electric or electronic implants, e.g. heart pacer
* any metal artefacts in the head
* Epilepsy
* Auto-immune diseases in acute stage
* mental diseases, e.g. schizophrenia etc.
* diabetic retinopathy
* addictive diseases
* blood pressure above 160/100 mmHg
* instable or high level of intraocular pressure above 27 mmHg
* retinitis pigmentosa
* pathological nystagmus
* presence of an un-operated tumor or tumor relapse (patients with non-progressive tumor are eligible if study participation is recommended by medical authorities)
* focal findings in EEG or photosensitivity (patients with single seizure more than 10 yrs ago may participate)
* recurrent transitional ischemic attacks after stroke
* arteriosclerosis of large blood vessels with stenosis >75%
* severe coronary heart disease (CHD)
* unstable angina pectoris
* diabetes with blood glucose level > 9 mmol/l
* myocard infarct/ cardiomyopathy
* ventricular fibrillation
* risk of vascular thrombosis
* pregnant or breast-feeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
detection accuracy (%) in visual field measures over baseline | baseline to 8 weeks after stimulation
  visual stimuli detection accuracy in residual and absolutely defect visual field will be assessed using computer-based high resolution perimetry (HRP)

SECONDARY OUTCOMES:
detection accuracy (%) in the intact visual field over baseline | baseline to 8 weeks after stimulation
  visual stimuli detection accuracy in the intact visual field will be assessed using computer-based high resolution perimetry (HRP)
visual acuity (LogRAD) | baseline to 8 weeks after stimulation
EEG parameters | baseline to 8 weeks after stimulation
  entrainment of stimulation frequencies (EEG power spectra) and measures of functional connectivity
conventional perimetry | baseline to 8 weeks after stimulation
  visual fields obtained by static and kinetic perimetry (average threshold in db, average excentricity in degrees)
reaction time (ms) | baseline to 8 weeks after stimulation
  average reaction time in ms, measured by computer-based high resolution perimetry (HRP)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard A Sabel, Ph.D., Principal Investigator — Univ. of Magdeburg
Locations (1):
- Inst. f. Medical Psychology, Univ. of Magdeburg, Magdeburg, Germany

REFERENCES:
- [Derived] Raty S, Borrmann C, Granata G, Cardenas-Morales L, Schoenfeld A, Sailer M, Silvennoinen K, Holopainen J, De Rossi F, Antal A, Rossini PM, Tatlisumak T, Sabel BA. Non-invasive electrical brain stimulation for vision restoration after stroke: An exploratory randomized trial (REVIS). Restor Neurol Neurosci. 2021;39(3):221-235. doi: 10.3233/RNN-211198. PMID 34219679